CLINICAL TRIAL: NCT05727670
Title: Improving Orthodontic Treatment of Patients With Dental Retention
Brief Title: Treatment of Retentive Teeth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Treatment of Retentive Teeth
Keywords: dental retention; digital dentistry; surgical navigation template; 3D printing

STUDY DESIGN:
Intervention Model Description: At the first stage of our study, it is planned to examine patients aged 15-35 years. The examination will be carried out according to the scheme including the main (clarification of complaints, anamnesis collection, external examination, examination of the oral cavity and teeth) and additional examination methods (anthropometric examination of diagnostic models of dentition, cone-beam computed tomography of the head, orthopantomography, telerentgenography of the head, electrodontodiagnostics, determination of the area of occlusal contacts).
  At the second stage of our study, it is planned to sample the results with the division of patients into the main and control groups. The main group will include patients who will receive orthodontic treatment according to the method we have proposed. The control group will include patients whose treatment will be carried out according to the standard method
Masking Description: development of a method for the treatment of extension of s with acceleration of treatment time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- main group (Experimental): This group consists of patients with dental retention who will be treated using digital technologies and devices to create a place in the dentition
  Interventions: Procedure: exposure of the tooth crown

INTERVENTIONS:
Procedure: exposure of the tooth crown — surgical exposure of the crown of a retentive tooth

SUMMARY:
The relevance of the research topic is beyond doubt, since this work is devoted to improving the effectiveness of treatment of patients with permanent teeth that have not erupted in a timely manner. Currently, this pathology occurs in 4-18% of patients seeking specialized help in a dental clinic.

The anomaly of teething, first of all, affects the anatomical, functional and aesthetic characteristics, there is an influence on the psycho-emotional state of the patient. Despite a significant number of scientific studies by domestic and foreign authors, some features of the treatment of patients with dental retention are insufficiently covered and systematized. At the moment, there is no optimal approach to the diagnosis and treatment of dental retention, as a result of which there is a question of improving the effectiveness and quality of orthodontic treatment of patients with a diagnosis of "tooth retention".

DETAILED DESCRIPTION:
The purpose of the study Improving the effectiveness of treatment of patients with dental retention. Research objectives

1. To determine the frequency of occurrence of dental retention according to the patients' requests for orthodontic care;
2. Based on the cephalometric study to identify the features of the structure of the face and bone structures in patients with dental retention;
3. Develop and implement an orthodontic device to obtain additional space in the dentition in patients with retention;
4. To develop and introduce into clinical practice a method for creating surgical access to retentive teeth using digital technologies.
5. To conduct a comparative analysis of the effectiveness of our proposed improved stages of treatment of patients with dental retention with well-known methods based on gnatic and profilometric indicators.

Materials and methods of research At the first stage of our study, it is planned to examine patients aged 15-35 years who have applied for specialized

ELIGIBILITY:
Inclusion Criteria:

* Methodology

Exclusion Criteria:

* patients without retentive teeth

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
treatment time | two years
  acceleration of treatment terms

CONTACTS AND LOCATIONS:
Locations (1):
- Irina, Samara, Samara Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
The orthodontic design developed by us will allow to create an additional place in the dentition with the subsequent extension of the retented tooth.
  The introduction into the clinical stage of the method we have developed for creating surgical access will facilitate the operation process and the number of complications.
Supporting Information: Study Protocol, CSR
Time Frame: three years